CLINICAL TRIAL: NCT05015114
Title: Prevalence and Factors of Sarcopenia in Patients With Primary Sjogren's Syndrome
Brief Title: Prevalence and Factors of Sarcopenia and in Patients With Primary Sjogren's Syndrome
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Özgül Öztürk, Assistant Professor, Acibadem University
Other Study IDs: ATADEK - 2021/10
Record Dates: First submitted 2021-08-12; First posted 2021-08-20 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Sarcopenia; Sjogren's Syndrome; Rheumatologic Disease
MeSH Terms: conditions — Sarcopenia; Sjogren's Syndrome; Collagen Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Sjogren's Syndrome: Participants with Primary Sjogren's Syndrome
  Interventions: Other: Sarcopenia Assessment
- Control group: Healthy controls
  Interventions: Other: Sarcopenia Assessment

INTERVENTIONS:
Other: Sarcopenia Assessment — Sarcopenia Assessment

SUMMARY:
Sarcopenia is a progressive condition characterized by decline in muscle strength and muscle mass. Although the mechanism of sarcopenia has not been fully elucidated, it may be caused by protein-poor diet, vitamin D deficiency, hormonal changes, increase in inflammatory cytokine level and oxidative stress. For this reason, it is thought that determining the prevalence of sarcopenia in rheumatological diseases with chronic inflammation and protecting patients from possible comorbidities with appropriate interventions may be an important factor in maintaining and improving the functional levels and quality of life of patients.

The aim of our study was to investigate the prevalence and its associated factors of sarcopenia in individuals with primary Sjögren's Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary Sjogren's syndrome by an experienced rheumatologist according to European League Against Rheumatism (EULAR) ve American College of Rheumatology (ACR) criteria
* Being 40 years or older.

Exclusion Criteria:

* Pregnancy,
* Malignancy,
* Presence of other rheumatological diseases,
* Presence of diabetes mellitus
* Presence of neurological problems
* Presence of osteoarthritis

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with primary Sjogren's syndrome
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Muscle Mass | 1 day
  Muscle mass will be calculated via bioimpedance analysis method. Fat Free Mass will be recorded using TANITA BC 532 Bioimpedance Device and Skeletal Muscle Mass and Skeletal Muscle Mass will be calculated.
Grip Strength | 1 day
  Grip strength will be evaluated with JAMAR dynamometer. The patient is positioned in a chair with the elbow flexed to 90 degrees and the wrist in a neutral position, and he/she is asked to grip as strong as he/she can do for 3 seconds. The test is repeated 3 times and the highest value is recorded.
Gait Speed | 1 day
  The patient will be asked to walk 4-meters for two times. The shortest time to walk through this distance will be recorded.
5 Times Sit to Stand Test | 1 day
  This test includes the calculation of the time it takes to sit and get up from the chair 5 times while the arms are crossed over the shoulders.

SECONDARY OUTCOMES:
EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) | 1 day
  ESSDAI was developed to determine the disease activity level specifically for Sjogren's Syndrome. It includes 12 domains (ie, organ systems: cutaneous, respiratory, renal, articular, muscular, peripheral nervous system (PNS), central nervous system (CNS), haematological, glandular, constitutional, lymphadenopathic, biological). Each domain is divided into 3-4 levels of activity. A score less than 5 indicates a low level of disease, a score between 5 and 13 indicates a moderate level, and a score of more than 14 indicates a high level of active 14. It is a scoring system that evaluates every domain between 0 and 3.
EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) | 1 day
  The patient is asked to define the level of fatigue, pain and dryness symptoms with a score between 1 and 10, and the average of the score obtained from these three questions are recorded. An ESSPRI score of less than 5 was considered an acceptable disease state, while a score of 5 or above was considered a sign of high activity.
Malnutrition Evaluation | 1 day
  The presence of malnutrition in the participants will be evaluated with the Mini Nutritional Assessment Form (Short Form). This form consists of 6 questions including loss of appetite, weight loss, mobility, stress or acute illness, dementia or depression, and body mass index. The total score ranges from 0 to 14, with 12 and above meaning "normal nutritional status", 8 to 11 "malnutrition risk" and 0 to 7 meaning malnutrition.

CONTACTS AND LOCATIONS:
Locations (1):
- Haydarpasa Numune Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No